CLINICAL TRIAL: NCT04349475
Title: Pilot RCT Intervention Targeting Elevated Triglycerides With a Point-of-Care Meter and Omega-3 Fatty Acids to Normalize Triglycerides and Fetal Growth
Brief Title: Therapeutic Omegas for Triglyceride Suppression
Acronym: TOTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-0707
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Pregnancy
Keywords: triglycerides; glucose; adiposity; Air displacement plethysmography; Continuous glucose monitoring
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega 3 Supplementation (Experimental): Supplementation of 4g of DHA/EPA daily
  Interventions: Dietary Supplement: Intervention Omega 3 Supplementation
- Safflower Oil Supplement (Placebo Comparator): Supplementation of Safflower Oil daily
  Interventions: Dietary Supplement: Control Safflower Oil

INTERVENTIONS:
Dietary Supplement: Intervention Omega 3 Supplementation — Participants will supplement 4g of Omega 3 fish oil daily (750DHA/250EPA)
  Arms: Omega 3 Supplementation
Dietary Supplement: Control Safflower Oil — Participants will consume 2.5g of a Safflower oil supplement daily
  Arms: Safflower Oil Supplement

SUMMARY:
This study plans to learn more about how an omega-3 fatty acid supplement effects triglyceride levels in pregnancy. Triglycerides are a type of fat found in your blood. Your body converts extra calories into triglycerides to be stored and used later for energy. It is normal for triglyceride levels to go up during pregnancy however some women have levels that are ~30-40% higher than normal when they reach their third trimester of pregnancy. Having high triglycerides in pregnancy may be related to an increased chance of having a baby that is large for their age. The goal of this study is to determine if taking an omega-3 fatty acid supplement can slow the rise in triglyceride levels later in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 21-39 yrs
* Pre-pregnancy BMI 28-39
* Fasting Triglyceride ≥120 mg/dL measured by 15 wks

Exclusion Criteria:

* Pre-gestational diabetes or prediabetes
* History of gestational diabetes,
* History of pre-eclampsia, spontaneous pre-term delivery, or gestational hypertension <34wks
* Tobacco or illicit substance use
* Chronic steroid use

Ages: 0 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal Fasting and Postprandial Triglycerides | 34 weeks gestational age
  Differences in maternal fasting and postprandial triglycerides between groups

CONTACTS AND LOCATIONS:
Overall Officials: Teri L Hernandez, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado/Anschutz Medical Campus, Aurora, Colorado
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

REFERENCES:
- [Background] Barbour LA, Farabi SS, Friedman JE, Hirsch NM, Reece MS, Van Pelt RE, Hernandez TL. Postprandial Triglycerides Predict Newborn Fat More Strongly than Glucose in Women with Obesity in Early Pregnancy. Obesity (Silver Spring). 2018 Aug;26(8):1347-1356. doi: 10.1002/oby.22246. Epub 2018 Jun 22. PMID 29931812